CLINICAL TRIAL: NCT07334288
Title: Efficacy of Ultrasound-Guided Retrolaminar Block Combined With Standard Multimodal Analgesia for Postoperative Pain Management in Lumbar Spine Surgery: A Randomized Controlled Trial
Brief Title: Retrolaminar Analgesia for LuMbar Surgery
Acronym: REALM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Nicolás Valls, Anesthesiologyst, Anesthesiology Department, Clínica Universidad de Los Andes, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUA2025-42
Record Dates: First submitted 2025-11-13; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Lumbar Surgery; Back Pain Lower Back Chronic; Opioid Analgesia; Regional Anaesthesia
Keywords: retrolaminar block; regional anesthesia; lumbar spine surgery; Multimodal analgesia; opioid consumption; Ultrasound-guided nerve block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Assignment, Blinded outcome assessment
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors (including pain evaluators and data collectors) will be blinded to group allocation.
  The anesthesiologist performing the intervention and the patient cannot be blinded due to the nature of the procedure (performance of nerve block).
  Postoperative care providers will also be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar Block & Standard Analgesia (Experimental): Patients receive bilateral ultrasound-guided retrolaminar blocks with Bupivacaine 0.25% and Epinephrine 50mcg (15 ml total volume per side) before surgery, along with standard multimodal analgesia.
  Interventions: Procedure: Ultrasound-Guided Retrolaminar Block
- Standard Analgesia Only (Active Comparator): Patients receive standard multimodal analgesia without regional anesthesia block.
  Interventions: Other: Standard Analgesia

INTERVENTIONS:
Procedure: Ultrasound-Guided Retrolaminar Block — Patients will receive bilateral ultrasound-guided retrolaminar blocks with Bupivacaine 0.25% and Epinephrine 50mcg (15 ml total volume per side) before surgery. The block will be performed by an experienced anesthesiologist using real-time ultrasound guidance.
  Arms: Retrolaminar Block & Standard Analgesia
Other: Standard Analgesia — Patients receive standard multimodal analgesia without regional anesthesia block.
  Arms: Standard Analgesia Only

SUMMARY:
This randomized controlled trial evaluates the effectiveness of ultrasound-guided retrolaminar nerve block in addition to standard multimodal analgesia for postoperative pain management in patients undergoing lumbar spine surgery. Fifty patients will be randomly assigned to receive either the retrolaminar block combined with standard pain management or standard pain management alone. The primary outcome is total opioid consumption in the first 24 hours after surgery. Secondary outcomes include pain intensity at multiple time points, time to first rescue analgesia, duration of sensory block, incidence of postoperative nausea and vomiting, length of hospital stay, patient satisfaction, and chronic pain development at 3 and 6 months follow-up.

DETAILED DESCRIPTION:
BACKGROUND: Lumbar spine surgery is associated with significant postoperative pain, which can delay recovery and increase complications. Regional anesthesia techniques, specifically retrolaminar blocks, may provide superior analgesia compared to systemic opioids alone.

STUDY DESIGN: This is a prospective, randomized, controlled trial conducted at Clínica Universidad de Los Andes, Chile. Patients will be allocated using variable block randomization (block sizes 4 and 6) in a 1:1 ratio.

INTERVENTIONS: All patients will receive standardized general anesthesia (Propofol, Remifentanil, Rocuronium) and multimodal analgesia including paracetamol, metamizol, ketorolac, morphine, and pregabalin. The intervention group will additionally receive bilateral ultrasound-guided retrolaminar blocks with ropivacaine 0.5% (20 ml per side) at the end of surgery.

OUTCOMES: Primary outcome is cumulative morphine consumption via patient-controlled analgesia (PCA) during the first 24 postoperative hours. Secondary outcomes include pain scores (VAS 0-10) at 0, 6, 12, 24, 48, and 72 hours; time to first rescue analgesia; duration of sensory block; incidence of nausea/vomiting; hospital length of stay; time to ambulation; sleep quality; patient satisfaction; adverse events; and development of chronic pain at 3 and 6 months.

SAMPLE SIZE: 50 patients (25 per group) provides 80% power to detect a clinically significant difference in opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-80 years
* Scheduled for elective lumbar spine surgery (with instrumentation)
* American Society of Anesthesiologists (ASA) physical status I-III
* Willing and able to provide written informed consent
* Able to use patient-controlled analgesia (PCA) device

Exclusion Criteria:

* Refusal to participate in the study
* Known allergy to local anesthetics (bupivacaine - levobupivacaine - lidocaine) or any study medication
* Contraindication to regional anesthesia (infection at injection site, coagulopathy)
* Chronic opioid use (daily use for >3 months prior to surgery)
* Severe psychiatric disorder that precludes informed consent
* Emergency surgery
* Diabetes mellitus with preoperative glucose >180 mg/dl
* Pregnancy or breastfeeding
* Body mass index (BMI) >40 kg/m²
* Reoperation or revision of the same level of previous spinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Total postoperative opioid consumption | First 24 hours after surgery
  Cumulative morphine consumption (in mg morphine equivalents) delivered via patient-controlled analgesia (PCA) pump during the first 24 postoperative hours

SECONDARY OUTCOMES:
Pain Intensity | Time in minutes from end of surgery until first request for rescue analgesia Time Frame: From end of surgery up to 72 hours
  Pain intensity measured using Visual Analog Scale (VAS, 0-10 where 0=no pain and 10=worst imaginable pain) Time Frame: 0, 6, 12, 24, 48, and 72 hours postoperatively
Duration of Sensory Block | From block performance up to 72 hours
  Duration in hours from block performance until complete sensory recovery assessed by thermal and tactile testing
Time to First Rescue Analgesia | From end of surgery up to 24 hours
  Time in minutes from end of surgery until first request for rescue analgesia
Incidence of PONV | First 24 hours postoperatively
  Incidence of postoperative nausea and vomiting (PONV) requiring antiemetic rescue medication
Length of hospital stay | From admission to discharge, assessed up to 30 days
  Total number of days from hospital admission to discharge

OTHER OUTCOMES:
Patient satisfaction | 72 hours postoperatively
  Patient satisfaction with pain management measured using 5-point Likert scale (1=very dissatisfied to 5=very satisfied)
Chronic Pain Development | 3 months and 6 months postoperatively
  Incidence of chronic pain defined as VAS > 3 at surgical site

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas J Valls, M.D, Ph.D, Study Director — Anesthesiologyst, Clinica Universidad de los Andes
Locations (1):
- Clínica Universidad de los Andes, Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification, will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available beginning 6 months and ending 5 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for use in achieving the aims of the approved proposal. Proposals should be directed to rcoloma@clinicauandes.cl. To gain access, data requestors will need to sign a data access agreement. Data will be shared after approval by the principal investigator and the institutional review board.

REFERENCES:
- [Background] Zeballos JL, Voscopoulos C, Kapottos M, Janfaza D, Vlassakov K. Ultrasound-guided retrolaminar paravertebral block. Anaesthesia. 2013 Jun;68(6):649-51. doi: 10.1111/anae.12296. No abstract available. PMID 23662765
- [Background] Ardon AE, Prasad A, McClain RL, Melton MS, Nielsen KC, Greengrass R. Regional Anesthesia for Ambulatory Anesthesiologists. Anesthesiol Clin. 2019 Jun;37(2):265-287. doi: 10.1016/j.anclin.2019.01.005. Epub 2019 Mar 15. PMID 31047129
- [Background] Batra RK, Krishnan K, Agarwal A. Paravertebral block. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):5-11. No abstract available. PMID 21804697
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT07334288/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT07334288/ICF_001.pdf